CLINICAL TRIAL: NCT02887911
Title: Characterization of Adults for Asthma Microbiome Research Studies (CAARS)
Brief Title: Characterization of Adults for Asthma Microbiome Research Studies
Acronym: CAARS
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Yvonne J Huang, Associate Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00097163; 5R01AI129958 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Asthma; Healthy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen samples will be retained indefinitely in a coded manner. It is anticipated that samples from this research study will be used in future research projects.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Asthmatic, not taking inhaled steroids: Men/Women, ages 18-75 who are not currently taking corticosteroids.. No intervention; this is a prospective observational study.
- Asthmatic, taking inhaled steroids: Men/Women, ages 18-75 who are already taking corticosteroids prescribed by their physician. No intervention; this is a prospective observational study.
- Healthy, non-asthmatic without allergies: Men/Women, ages 18-75 without a current diagnosis of asthma and no allergies. No intervention; this is a prospective observational study.
- Healthy, atopic non-asthmatic: Men/Women, ages 18-75 with allergies but without a current diagnosis of asthma. No intervention; this is a prospective observational study.

SUMMARY:
The purpose of this study is to characterize adult subjects regarding their history of allergy and asthma, clinical manifestations of asthma, and exposures and conditions that may influence asthma severity and control. Assessments include baseline medical history, lung function tests, questionnaires, and collection of specimens for phenotypic characterization.

DETAILED DESCRIPTION:
This is a prospective, observational study in which approximately 200 subjects will be enrolled, including healthy controls, atopic controls without asthma, and patients with stable asthma (n = 150). Among asthmatics, 2/3 will be on regular inhaled corticosteroid therapy and 1/3 will not be taking inhaled corticosteroids. Subjects who meet study criteria will undergo phenotypic characterization in multiple domains, including evaluation of lung function, assessments of asthma/allergy history, asthma triggers, asthma symptom control, environmental microbial exposures and dietary intake. Oral rinse, sputum, stool, urine and blood specimens will be collected for microbiome-related analyses, including molecular and culture-based assays, metabolite studies, and to relate these to markers of inflammation and immune function. The overall goal is to enroll a cohort of well-characterized asthmatic and non-asthmatic control subjects to enable mechanism-oriented studies of how members of the airway microbiota and possibly also gut microbiota influence phenotypes of adult asthma.

ELIGIBILITY:
1. For all subjects:

   Inclusion criteria:

   - Men/Women, ages 18-75, with or without current asthma, are eligible to be screened.

   Exclusion criteria:
   * Cigarette smoking history of >30 total pack-years
   * Current use of other smoked products or recreational drugs (e.g. pipes, cigars, e-cigarettes, other illicit drugs)
   * History of lung disease other than asthma
   * Recent upper respiratory tract infection treated with antibiotics within 8 weeks of visit 1
   * Recent antibiotic use (except topical or ocular) within 8 weeks of visit 1 (chronic antibiotic use for asthma management allowed)
   * Currently pregnant or breast-feeding
   * Other medical conditions or treatments that may increase subject risk or affect study results, based on study physician judgment. These include the following: significant cardiovascular disease(+/- active symptoms), arrhythmia, or stroke, active cancer, post-organ transplant
   * Any other condition for which subject is taking immunosuppressive therapies (except steroids for asthma)
   * History of allergy to albuterol or methacholine
2. For asthma subjects only:

   Note: Enrollment target is for 90 asthmatics already taking inhaled corticosteroids prescribed by their physician (any formulation and dose) and 60 subjects who are not currently using inhaled corticosteroid.

   Additional inclusion criteria:
   * History of asthma symptoms within the last 2 years (e.g. wheeze, shortness of breath, etc.)
   * Evidence of stable asthma as assessed by initial screening
   * No changes in asthma medications within 30 days of visit 1
   * Methacholine PC20 (dose at which there is a 20 percent change) ≤ 8 mg/ml (for those asthmatics on inhaled steroids, PC20 ≤ 16 mg/ml), or change in FEV1 (forced expiratory volume in first second of spirometry effort)≥ 12% after 4 puffs of albuterol on reversibility testing (or PI discretion)
   * If negative methacholine challenge or no evidence of bronchodilator reversibility, a strong history of physician-diagnosed/physician-managed asthma may allow for study inclusion, based on PI's judgement or discretion.
   * Individuals with a history of physician-diagnosed asthma who have had bronchodilator reversibility testing or methacholine challenge performed within 60 days of screening may be enrolled and these existing test results used in lieu of repeating the same test at visit 1 or visit 2.

   Additional exclusion criteria:
   * An asthma exacerbation requiring treatment with oral or IV steroids within 1 month of visit 1
   * No asthma symptoms within the last 2 years
3. For healthy control or atopic non-asthma subjects:

Additional exclusion criteria:

* Evidence of abnormal lung function by any of the following: FEV1/FVC ratio <0.70, FEV1 or FVC (forced vital capacity on spirometry) < 80% predicted, methacholine PC20 < 16 mg/ml, or FEV1 improvement > 12% in response to albuterol
* Atopic non-asthma subjects found to have evidence of abnormal lung function, but without a clear or recent history of asthma, may be enrolled per PI's discretion.
* Possible pulmonary disease is identified by PI or Co-Is to explain an abnormal lung function result at the time of testing. The subject may be re-screened later at investigator's discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of well characterized asthmatic subjects and a cohort of healthy people without asthma.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
To characterize adult subjects with asthma in multiple domains, including disease severity and control, patterns of airway inflammation, microbial exposures and patterns of airway and gut microbial colonization | Day 1" for the first one and "up to 60 days"

SECONDARY OUTCOMES:
To evaluate differences in airway and gut microbiota composition related to inhaled corticosteroid use (ICS) among asthmatics already regularly taking ICS, asthmatics not taking ICS, and healthy controls | Day 1" for the first one and "up to 60 days"

OTHER OUTCOMES:
To apply culture and molecular methods to study functions of asthma-associated airway microbiota in corticosteroid-enriched environments | Day 1" for the first one and "up to 60 days"
To evaluate the temporal stability of the airway microbiome in asthmatic and healthy subjects | Day 1" for the first one and "up to 60 days"
To explore relationships between airway and gut microbiome composition in asthma, including among obese subjects | Day 1" for the first one and "up to 60 days"

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne J. Huang, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No